CLINICAL TRIAL: NCT01241643
Title: A Multicenter, Open-labeled, Controlled, Randomized Study of Recombinant Interleukin-7 (CYT107) Treatment to Restore and Maintain CD4 T-lymphocyte Counts Above 500 Cells/µL in HIV-infected Patients With CD4 Counts Remaining Between 101-350 Cells/µL After at Least 2 Years of HAART and Plasma HIV RNA < 50 Copies/mL for 18 Months.
Brief Title: Randomized Study on Multiple Cycles of Interleukin-7 in HIV Patients Immune Non-responders
Acronym: Inspire 3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated [CYTHERISSA filed for banckcuptcy in June 2013.Subjects treated by CYT107 were followed up for at the least 3 months.]
Sponsor: Cytheris SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLI-107-14
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: HIV
Keywords: interleukin-7; immune-based therapies; HIV; infectious disease; immune non-responders
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYT107 (Experimental): repeated cycles of CYT107 at 20 µg/kg/week over 2 weeks, for a maximum of 4 cycles within 21 months and a maximum of 3 cycles within 12 months
  Interventions: Drug: CYT107
- Control (No Intervention): Control arm with possible CYT107 injection after 12 months of study participation

INTERVENTIONS:
Drug: CYT107 — repeated cycles of 3 injections of CYT107 at 20 µg/kg/week over 2 weeks, for a maximum of 4 cycles within 21 months and a maximum of 3 cycles within 12 months
  Arms: CYT107

SUMMARY:
This is a Phase II multicenter, open-labeled, controlled, randomized study assessing weekly doses of Interleukin-7 (CYT107)

DETAILED DESCRIPTION:
The aim of the study is to assess repeated cycles of 3 weekly injections of CYT107 in patients immune non-responders infected with HIV.

Eighty patients will be recruited to study the biological activity and safety of repeated cycles of CYT107 at 20 µg/kg/week over 2 weeks, for a maximum of 4 cycles within 21 months and a maximum of 3 cycles within 12 months. The entire study will cover a period of 24 months.

During the study visits the following may be done:

* medical history, physical examination, blood test every visit
* EKG
* chest X-Ray
* liver/spleen ultrasound

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection as documented by any licensed ELISA (Enzyme-Linked Immunosorbent Assay) test kit and confirmed either by Western Blot or a 2nd test using a different method at any time prior to study entry
2. Age ≥18
3. On HAART (Highly active anti-retroviral therapy) for at least 24 months, on stable regimen for at least 6 months prior to study entry. HAART is defined as a combination of two (2) classes dose regimen of approved ARV (antiretroviral)
4. CD4+ cell counts ≥ 101 and < 350 cells/µL measured on at least two (2) measurements (including the screening value) within the previous 12 months prior to study entry Note: a single isolated value of CD4+ ≥ 350 during this period (12 months prior to study entry) will be allowed to participate if the previous and subsequent CD4+ count is in the range of ≥ 101 and < 350 cells/µL
5. Plasma HIV RNA < 50 copies/mL since at least 18 months with at least two (2) measurements (including the screening value) within the previous 6 months prior study entry Note: patients with single blip of detectable viremia during this period (6 months prior to study entry) will be allowed to participate if the prior and subsequent plasma HIV RNA levels are < 50 copies/mL
6. Adequate bone marrow, hepatic and renal function as follows:

   * Hemoglobin ≥ 10 g/dl
   * Neutrophils ≥ 1,000/µL
   * Platelets ≥ 100,000/µL
   * AST, ALT, or Alk. Phosph. ≤ 2.5 x ULN
   * Total Bilirubin ≤ 1.5 x ULN (or ≤ 5 x ULN if the patient is treated by atazanavir or by indinavir, and if the increase is due to unconjugated bilirubin and if ALT and AST are normal)
   * Lipase ≤ 2 x ULN
   * PT/PTT ≤ 1.5 x ULN
   * Estimated glomerular filtration ≥ 60 ml/min (according to MDRD formula)
7. Normal blood Thyroid-Stimulating Hormone (TSH)
8. Ability to understand and sign informed consent

Exclusion Criteria:

1. AIDS-defining illness (category C) diagnosed within the last 12 months prior to study entry
2. History of HIV related encephalopathy
3. Active opportunistic infection including active tuberculosis
4. Previous treatment with IL-2 or IL-7 at any time prior to study entry
5. Any planned or probable modification of the anti-retroviral treatment during the first year or the first two cycles of CYT107 Note: in case of product shortage and in absence of viral mutation suspicion or viral blip, a modification of ARV will not be an exclusion criterion
6. Poor compliance on HAART or any other chronic treatment that in the opinion of the investigator will interfere with protocol participation
7. Previous treatment with immuno-modulatory agents such as, systemic corticosteroids, growth factors, immunosuppressive drugs, HIV vaccine, or anti-cancer treatment or hydroxyurea within 3 months prior to study entry
8. Any history of malignancy (except basal carcinoma of the skin) including any hematologic malignancy or AIDS defining malignancy, such as lymphoproliferative disorder or Kaposi's sarcoma Note: Patients with Kaposi's sarcoma limited to the skin that had disappeared while on HAART therapy, and without requiring any other systemic therapy 1 year prior to study entry, will be eligible.
9. Any history of severe auto-immune disease requiring systemic treatment or hospitalization, or any active auto-immune disease requiring treatment (including multiple sclerosis)
10. History of splenectomy
11. Any hematologic disease associated with hypersplenism, such as thalassemia, hereditary spherocytosis, Gaucher's Disease, and autoimmune hemolytic anemia
12. Chronic hepatitis B or C
13. HIV-2, HTLV-1 or HTLV-2 seropositivity
14. Cirrhosis of any origin, and alcoholic or non alcoholic steato-hepatitis, either proven histologically or suspected
15. Hypertension with a resting systolic blood pressure > 140 or a resting diastolic blood pressure > 90 mm despite adequate antihypertensive treatment
16. Any cardiac, pulmonary, thyroid, renal, hepatic, gastrointestinal, neurological (central or peripheral) disease requiring therapy and considered as significant by the investigator or a severe disorder of hemostasis
17. Any serious illness requiring systemic treatment and/or hospitalization until the patient either completes therapy or is clinically stable on therapy, in the opinion of the principal investigator, for at least 30 days prior to study entry
18. Pregnant or lactating women. Women of childbearing potential must have a negative serum or urine pregnancy test at study entry
19. Refusal or inability to practice contraception regardless of the gender of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To study the biological activity and safety of repeated cycles of CYT107 at 20 µg/kg/week over 2 weeks, for a maximum of 4 cycles within 21 months and a maximum of 3 cycles within 12 months. | 24 months

SECONDARY OUTCOMES:
To characterize CYT107 Pharmacokinetics (PK) / Pharmacodynamics (PD) | 24 months
To characterize the key immuno-pharmacological effects | 24 months
To assess CYT107 effect on HIV-induced chronic systemic immune hyper-activation and its consequences | 24 months

CONTACTS AND LOCATIONS:
Locations (3):
- San Raffaele Scientific Institute, Milan, Italy
- Helen Joseph Hospital-Themba Lethu Clinic, Johannesburg, South Africa
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Thiebaut R, Jarne A, Routy JP, Sereti I, Fischl M, Ive P, Speck RF, D'Offizi G, Casari S, Commenges D, Foulkes S, Natarajan V, Croughs T, Delfraissy JF, Tambussi G, Levy Y, Lederman MM. Repeated Cycles of Recombinant Human Interleukin 7 in HIV-Infected Patients With Low CD4 T-Cell Reconstitution on Antiretroviral Therapy: Results of 2 Phase II Multicenter Studies. Clin Infect Dis. 2016 May 1;62(9):1178-1185. doi: 10.1093/cid/ciw065. Epub 2016 Feb 7. PMID 26908786